CLINICAL TRIAL: NCT00005262
Title: Epidemiology of Idiopathic Dilated Cardiomyopathy (Washington, DC Dilated Cardiomyopathy Study)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1146; R29HL044904 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Diseases; Asthma; Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Cardiomyopathies; Asthma; Diabetes Mellitus; Hypertension

SUMMARY:
To identify risk factors for idiopathic dilated cardiomyopathy and to examine prognostic factors over a follow-up period of two to three years.

DETAILED DESCRIPTION:
BACKGROUND:

Idiopathic dilated cardiomyopathy is an often fatal cause of heart failure in young adults which is characterized by dilatation of the ventricles, increased myocardial mass, and impairment of systolic function. Dilated cardiomyopathy is more common than hypertrophic and restrictive cardiomyopathy, and the symptoms and physical signs are those of left-sided and eventually right-sided heart failure. Histologic findings in the condition include nonspecific interstitial myocardial fibrosis and myocyte hypertrophy. Despite the large number of systemic or generalized disease processes which have been associated with secondary dilated cardiomyopathy, the majority of cases are idiopathic. Mortality rates from cardiomyopathy have increased dramatically since 1970, and in 1990 over 10,000 deaths annually were attributed to cardiomyopathy in the United States.

DESIGN NARRATIVE:

The study had a prospective case-control design. Medical records of possible cases of idiopathic dilated cardiomyopathy who were discharged from five Washington, D. C. acute care hospitals over a two year period were abstracted so that standard diagnostic criteria could be applied. Two neighborhood controls were identified for each case. Cases and controls were matched on five year age intervals, sex, and telephone exchange. Cases were contacted annually during the two to three year follow-up period to determine vital status. The study determined whether the reported association between idiopathic dilated cardiomyopathy and asthma could be confirmed and the possible role of asthma medications, cigarette smoking, moderate alcohol consumption, and diabetes mellitus in the etiology of idiopathic dilated cardiomyopathy. The role of hypertension was also studied.. Statistical analysis consisted of case-control comparisons using conditional logistic regression techniques, and survival analyses using Kaplan-Meier curves and proportional hazards models.

The study was also known as the Washington, D.C. Dilated Cardiomyopathy Study. Dr. Coughlin started his research at Georgetown University in Washington, D.C. and transferred to Tulane University.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-07; Study Completion 1996-06 (Actual)

REFERENCES:
- [Background] Coughlin SS, Myers L, Michaels RK. What explains black-white differences in survival in idiopathic dilated cardiomyopathy? The Washington, DC, Dilated Cardiomyopathy Study. J Natl Med Assoc. 1997 Apr;89(4):277-82. PMID 9145633
- [Background] Metayer C, Coughlin SS, Mather FJ. Does cigarette smoking paradoxically increase survival in idiopathic dilated cardiomyopathy?. The Washington, D.C., Dilated Cardiomyopathy Study. Cardiology. 1996 Nov-Dec;87(6):502-8. doi: 10.1159/000177146. PMID 8904678
- [Background] Coughlin SS, Rice JC. Obesity and idiopathic dilated cardiomyopathy. Epidemiology. 1996 Nov;7(6):629-32. doi: 10.1097/00001648-199611000-00011. PMID 8899390
- [Background] Coughlin SS, Tefft MC, Rice JC, Gerone JL, Baughman KL. Epidemiology of idiopathic dilated cardiomyopathy in the elderly: pooled results from two case-control studies. Am J Epidemiol. 1996 May 1;143(9):881-8. doi: 10.1093/oxfordjournals.aje.a008831. PMID 8610701
- [Background] Coughlin SS, Pickle LW, Goodman MT, Wilkens LR. The logistic modeling of interobserver agreement. J Clin Epidemiol. 1992 Nov;45(11):1237-41. doi: 10.1016/0895-4356(92)90164-i. PMID 1432004
- [Background] Coughlin SS, Beauchamp TL. Ethics, scientific validity, and the design of epidemiologic studies. Epidemiology. 1992 Jul;3(4):343-7. doi: 10.1097/00001648-199207000-00009. PMID 1637897
- [Background] Coughlin SS, Pickle LW. Sensitivity and specificity-like measures of the validity of a diagnostic test that are corrected for chance agreement. Epidemiology. 1992 Mar;3(2):178-81. doi: 10.1097/00001648-199203000-00017. PMID 1576224
- [Background] Coughlin SS, Trock B, Criqui MH, Pickle LW, Browner D, Tefft MC. The logistic modeling of sensitivity, specificity, and predictive value of a diagnostic test. J Clin Epidemiol. 1992 Jan;45(1):1-7. doi: 10.1016/0895-4356(92)90180-u. PMID 1738006
- [Background] Coughlin SS, Nass CC, Pickle LW, Trock B, Bunin G. Regression methods for estimating attributable risk in population-based case-control studies: a comparison of additive and multiplicative models. Am J Epidemiol. 1991 Feb 1;133(3):305-13. doi: 10.1093/oxfordjournals.aje.a115875. PMID 2000848
- [Background] Coughlin SS, Chiazze L Jr. Job-exposure matrices in epidemiologic research and medical surveillance. Occup Med. 1990 Jul-Sep;5(3):633-46. PMID 2218806
- [Background] Coughlin SS, Metayer C, McCarthy EP, Mather FJ, Waldhorn RE, Gersh BJ, DuPraw S, Baughman KL. Respiratory illness, beta-agonists, and risk of idiopathic dilated cardiomyopathy. The Washington, DC, Dilated Cardiomyopathy Study. Am J Epidemiol. 1995 Aug 15;142(4):395-403. doi: 10.1093/oxfordjournals.aje.a117647. PMID 7625404
- [Background] Benton RE, Coughlin SS, Tefft MC. Predictors of coronary angiography in patients with idiopathic dilated cardiomyopathy: the Washington, DC Dilated Cardiomyopathy Study. J Clin Epidemiol. 1994 May;47(5):501-11. doi: 10.1016/0895-4356(94)90297-6. PMID 7730876
- [Background] Coughlin SS, Gottdiener JS, Baughman KL, Wasserman A, Marx ES, Tefft MC, Gersh BJ. Black-white differences in mortality in idiopathic dilated cardiomyopathy: the Washington, DC, dilated cardiomyopathy study. J Natl Med Assoc. 1994 Aug;86(8):583-91. PMID 7932836
- [Background] Coughlin SS, Tefft MC. The epidemiology of idiopathic dilated cardiomyopathy in women: the Washington DC Dilated Cardiomyopathy Study. Epidemiology. 1994 Jul;5(4):449-55. doi: 10.1097/00001648-199407000-00012. PMID 7918816
- [Background] Coughlin SS, Pearle DL, Baughman KL, Wasserman A, Tefft MC. Diabetes mellitus and risk of idiopathic dilated cardiomyopathy. The Washington, DC Dilated Cardiomyopathy Study. Ann Epidemiol. 1994 Jan;4(1):67-74. doi: 10.1016/1047-2797(94)90044-2. PMID 8205273
- [Background] Coughlin SS. A ban on policy recommendations in epidemiology research papers? Surely, you jest! Epidemiology. 1994 Mar;5(2):257-8. doi: 10.1097/00001648-199403000-00018. No abstract available. PMID 8173003
- [Background] Coughlin SS, Comstock GW, Baughman KL. Descriptive epidemiology of idiopathic dilated cardiomyopathy in Washington County, Maryland, 1975-1991. J Clin Epidemiol. 1993 Sep;46(9):1003-8. doi: 10.1016/0895-4356(93)90167-y. PMID 8263572
- [Background] Coughlin SS, Labenberg JR, Tefft MC. Black-white differences in idiopathic dilated cardiomyopathy: the Washington DC dilated Cardiomyopathy Study. Epidemiology. 1993 Mar;4(2):165-72. doi: 10.1097/00001648-199303000-00013. PMID 8452906
- [Background] Coughlin SS, Benichou J, Weed DL. Attributable risk estimation in case-control studies. Epidemiol Rev. 1994;16(1):51-64. doi: 10.1093/oxfordjournals.epirev.a036144. No abstract available. PMID 7925727
- [Background] Coughlin SS, Neaton JD, Sengupta A, Kuller LH. Predictors of mortality from idiopathic dilated cardiomyopathy in 356,222 men screened for the Multiple Risk Factor Intervention Trial. Am J Epidemiol. 1994 Jan 15;139(2):166-72. doi: 10.1093/oxfordjournals.aje.a116978. PMID 8296783